CLINICAL TRIAL: NCT04002232
Title: Prevention of Enamel Demineralization in Fixed Appliance Orthodontic Patients Using CPP-ACP-NaF Varnish Compared to Blank Varnish Base. A Randomized Split Mouth Controlled Clinical Trial
Brief Title: Prevention of Enamel Demineralization Using CPP-ACP-NaF Varnish
Acronym: CPP-ACP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-0968
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Demineralization

STUDY DESIGN:
Intervention Model Description: Split mouth
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo and the CPP-ACP-NaF varnishes will be supplied by the manufacturer labeled as either A or B. The blinding code is provided in a sealed envelop should there be a need to unblind the experiments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CPP-ACP-NaF (Experimental): Dental varnish that contains calcium phosphoprotein stabilized amorphous calcium phosphate and sodium fluoride (CPP-ACP-NaF) is applied to the teeth with orthodontic brackets on one side of the mouth immediately after the teeth have received the bracket.
  Interventions: Device: CPP-ACP-NaF varnish
- Placebo (Placebo Comparator): Dental varnish base that does not contain calcium phosphoprotein stabilized amorphous calcium phosphate and sodium fluoride (CPP-ACP-NaF) is applied to the teeth with orthodontic brackets on one side of the mouth immediately after the teeth have received the bracket.
  Interventions: Device: CPP-ACP-NaF varnish

INTERVENTIONS:
Device: CPP-ACP-NaF varnish — calcium phosphate containing fluoride releasing varnish to prevent caries

SUMMARY:
Sometimes when people wear braces, the combination of dental plaque and diets high in sugar and acids can lead to white spots on the teeth surrounding the braces. These are commonly found in people with braces depending on their diet and care of their teeth. The white spots will still be present when the braces are removed. These white spots are the beginning signs of cavities and show that mineral has been lost from the tooth. This study will be testing a new varnish that is painted on the tooth around the braces to prevent these white spots from forming.

This study will enroll patients who wear braces and have planned teeth extractions. A calcium and fluoride releasing varnish will be painted on the teeth planned to be extracted. Braces will then be placed on the teeth. In 3-6 weeks, the extraction will occur and the teeth will be collected for analysis.

DETAILED DESCRIPTION:
This is a randomized split mouth double blinded clinical trial. The CPP-ACP-NaF varnish is commercially available and is used for the treatment of tooth hypersensitivity under FDA 510K K102808. The placebo for this study is the same product without the CPP-ACP-NaF component. Patients with planned orthodontic therapy that include tooth extractions will have orthodontic brackets attached to the to-be-extracted teeth. Each patient will have the CPP-ACP-NaF varnish and the varnish base (without CPP-ACP-NaF) applied to teeth immediately after orthodontic brackets have been applied. The specific teeth (left or right) will be randomly determined as to the application of the varnish or placebo. In this experimental design each patient has CPP-ACP-NaF applied to one side and placebo applied to the other side.

When the teeth are extracted they are transferred to the Carey Laboratory for in vitro evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the University of Colorado School of Dental Medicine Department of Orthodontics who agree to consent to this study.
* Orthodontic treatment plans that include fixed appliances from the second premolar to second premolar in both arches.
* Orthodontic treatment plans that include extractions of at least 3 bicuspids for orthodontic therapy
* At least 10 years of age
* The patient has adequate oral hygiene

Exclusion Criteria:

* Evidence of decalcification or restorations on any of the premolars planned for extraction prior to orthodontic treatment
* Younger than 10 years of age
* Allergies to cow's milk or cow's milk products
* Any condition that contraindicates orthodontic treatment, or are not willing to consent to the study.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Demineralization | Up to 14 days after teeth extractions
  mineral density as determined by micro computed tomography (uCT)
Caries location | Up to14 days after teeth extractions
  Canary number that indicates early demineralization determined by the Canary System for caries identification

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Carey, Principal Investigator — University of Colorado, SoDM
Locations (1):
- University of Colorado School of Dental Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marinho VC, Higgins JP, Logan S, Sheiham A. Topical fluoride (toothpastes, mouthrinses, gels or varnishes) for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2003;2003(4):CD002782. doi: 10.1002/14651858.CD002782. PMID 14583954
- [Result] Nalbantgil D, Oztoprak MO, Cakan DG, Bozkurt K, Arun T. Prevention of demineralization around orthodontic brackets using two different fluoride varnishes. Eur J Dent. 2013 Jan;7(1):41-7. PMID 23408742
- [Result] Reynolds EC. Remineralization of enamel subsurface lesions by casein phosphopeptide-stabilized calcium phosphate solutions. J Dent Res. 1997 Sep;76(9):1587-95. doi: 10.1177/00220345970760091101. PMID 9294493
- [Result] Srivastava K, Tikku T, Khanna R, Sachan K. Risk factors and management of white spot lesions in orthodontics. J Orthod Sci. 2013 Apr;2(2):43-9. doi: 10.4103/2278-0203.115081. PMID 24987641
- [Result] Todd MA, Staley RN, Kanellis MJ, Donly KJ, Wefel JS. Effect of a fluoride varnish on demineralization adjacent to orthodontic brackets. Am J Orthod Dentofacial Orthop. 1999 Aug;116(2):159-67. doi: 10.1016/s0889-5406(99)70213-1. PMID 10434089